CLINICAL TRIAL: NCT04960241
Title: Physical Rehabilitation Versus no Physical Rehabilitation After Total Hip and Knee Arthroplasties: Protocol for a Pragmatic, Randomized, Controlled, Replication Trial (DRAW2)
Brief Title: Does Rehabilitation After Total Hip Or Knee Arthroplasty Work (DRAW2)
Acronym: DRAW2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Troels Mark Christensen (Other Government)
Responsible Party: Sponsor-Investigator, Troels Mark Christensen, Principal investigator, Bornholms Regionskommune
Organization: Bornholms Regionskommune (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Bornholms Regionskommune
Record Dates: First submitted 2021-07-02; First posted 2021-07-13 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2024-10

CONDITIONS: Rehabilitation; Telerehabilitation; Arthroplasty, Replacement, Hip; Arthroplasty, Replacement, Knee
Keywords: Rehabilitation; Telerehabilitation; No intervention; Total hip arthroplasty; Total knee arthroplasty

STUDY DESIGN:
Intervention Model Description: Homebased telerehabiltation. Homebased rehabilitation. No physical rehabilitation.
Who Masked: Care Provider, Outcomes Assessor
Masking Description: A physiotherapist will assess the outcomes at baseline after which the patients are randomized. The same physiotherapist will then deliver the allocated intervention and no longer assess outcomes for this patient. A different physiotherapist, who is blinded to treatment allocation, will assess outcomes at the follow-up visits in this patient. At all follow-up visits, patients will be asked not to disclose any information regarding group allocation, and the physiotherapists will be instructed not to ask questions regarding group allocation.
  The patients are blinded to the trial hypothesis in order to prevent ascertainment bias. The principal investigator is not an outcome assessor and will not be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Homebased telerehabilitation (Active Comparator): Patients randomized to this group will receive interactive virtual rehabilitation using a mobile app. The telerehabilitation is based on sensor technology, developed by ICURA. This technology consists of motion sensors that can measure and analyse the quantity and quality of the exercises, and a mobile application that can guide the patient with visual response. A unique feature of ICURA trainer allows the physiotherapist to remotely supervise the individual patients exercise adherence and progress. This technology has already been successfully implemented in several different rehabilitation facilities across Denmark, and, hence, reflects current clinical practice.
  Interventions: Procedure: Homebased telerehabilitation
- Homebased rehabilitation (Active Comparator): This group will be instructed in similar exercises as patients allocated to telerehabilitation. However, this group will receive a written exercise-program with instructions to perform these exercises at home. The home-based exercise program will be created using exercise templates from Exorlive. Using a link provided in the exercise-program, the patients will be able to see short instruction-videos of the individual exercises.
  Interventions: Procedure: Homebased rehabilitation
- No physical rehabilitation (Active Comparator): This group of randomised patients will not be given any physical rehabilitation intervention. This means no physical activity or exercise designed and prescribed for restoring normal function or reducing pain cause by disease, injury or surgery. The no intervention group will be encouraged to stay active and continue life as usual, gradually returning to their activities of daily living when they feel ready for it.
  Interventions: Procedure: No physical rehabilitation

INTERVENTIONS:
Procedure: Homebased telerehabilitation — The telerehabilitation intervention is based on sensor technology, developed by ICURA. The technology consists of motion sensors that can measure and analyse the quantity and quality of the exercises, and a mobile application that can guide the patients with visual response. A unique feature of ICURA trainer allows the physiotherapist to remotely supervise the individual patients exercise adherence and progress. The patients will receive a suitcase with five sensors (to be placed bilaterally on lower legs, thighs and one around the waist), a smartphone to record the exercises and a charging station free of charge during the 6-week intervention. At the end of the intervention the material will be returned at the first follow-up (t1). For more information please visit https://icura.dk.
  Arms: Homebased telerehabilitation
Procedure: Homebased rehabilitation — The unsupervised rehabilitation group will receive a written exercise program in order to perform daily exercises at home. The exercise program will be made using Exorlive (for more information about Exorlive please visit https://www.exorlive.com). In addition to the written program, patients will able to use a link provided to see small video-instructions on the internet of each exercise on the program. No feedback or supplementary instructions will be given after the initial face-to-face appointment.
  Arms: Homebased rehabilitation
Procedure: No physical rehabilitation — Patients allocated to the no intervention group will receive encouragement to stay active and be encouraged to gradually return to activities of daily living. This will be the only exercise-encouragement given to the no-intervention group.
  Arms: No physical rehabilitation

SUMMARY:
Overall frame: The overall or "parent" DRAW-project is a large-scale project run in Denmark that aims to provide substantial level 1A evidence-data related to the question: Does rehabilitation after total hip and knee replacements work? In the DRAW project, the authors challenge the belief that physical rehabilitation is clinically important - and surely better than "no physical rehabilitation". To challenge this belief thoroughly, the DRAW project holds many individual work packages centered around the same question. These work packages will be conducted in collaboration with municipality rehabilitation centers in Denmark so that specific usual care strategies are reflected in the different trials and local clinical relevance is as well as implementation potential are increased.

DETAILED DESCRIPTION:
The DRAW2-trial is a pragmatic, randomised controlled trial that aims to replicate the DRAW1-trial findings (clinicaltrials.gov: NCT03750448, trial protocol: https://f1000research.com/articles/10-146). Based on stakeholder input from Municipality Rehabilitation Bornholm, the DRAW1-trial was designed as a superiority trial to test the hypothesis that physical rehabilitation (telerehabilitation and home-based rehabilitation) is superior to no physical rehabilitation in a mixed population of patients after total hip and knee arthroplasty (THA and TKA, respectively). After DRAW1-trial inclusion was completed and the target sample size reached, an opportunity to continue the trial presented because additional funding was obtained. At the same time, Municipality Rehabilitation Bornholm asked for stratified data (THA/TKA) that could help guide their decision concerning a potential purchase of telerehabilitation equipment (more details on stakeholder input can be found in the trial protocol, https://f1000research.com/articles/10-146). To meet this new research objective of stratified analysis for THA and TKA, it was advised from the local ethical committee that a new and almost identical trial was registered, which would allow for a doubling of the sample simple size, so that adequately powered stratified analyses could be made. This new trial is named the DRAW2-trial.

The DRAW2-trial will adhere to the published DRAW1-trial protocol (https://f1000research.com/articles/10-146) and only small logistic modifications to trial procedures have been made. Because some of the DRAW1-trial participants felt overwhelmed by the amount of information they received during the first and only study introduction (usually takes place 5-7 days after surgery), the study introduction in the DRAW2-trial can be divided into two separate consultations a few days apart whenever deemed appropriate by the consulting physiotherapist. The DRAW2 trial will be reported and published independently, including the same outcomes and outcome hierarchy as the DRAW1-trial. As such, it will be an independent replication trial.

Research plan

While the DRAW2-trial will focus on replication of the DRAW-1 trial findings, the opportunity to run a replication trial at the same trial site with little delay between the two trials will also enable us to address the questions outlined below, by subsequent pooling of data from the two trials.

Question 1: Is physical rehabilitation superior to no physical rehabilitation after THA and TKA using two usual care strategies in Denmark (stratified analyses THA vs. TKA by pooling DRAW1 and 2 trial data)?

Question 2: Is home-based rehabilitation as good as home-based telerehabilitation in a mixed population of THA and TKA using two usual care strategies in Denmark (equivalence analysis by pooling DRAW1 and 2 trial data)?

Question 3: Is physical rehabilitation superior to no physical rehabilitation after THA in general (using DRAW1 and 2 THA trial data in an ongoing living systematic review? (https://www.crd.york.ac.uk/prospero/display_record.php?RecordID=203574).

Question 3: Is physical rehabilitation superior to no physical rehabilitation after TKA in general (using DRAW1 and 2 TKA trial data in an ongoing living systematic review? (https://www.crd.york.ac.uk/prospero/display_record.php?ID=CRD42018094785).

ELIGIBILITY:
Inclusion Criteria:

Patients having had primary, unilateral THA or TKA due to osteoarthritis. Patients being referred to receive postoperative rehabilitation at our institution.

Patients being able to speak, read and understand Danish language. Patients aged ≥ 18 years.

Exclusion Criteria:

Patients not able to comply with exercise instructions. Patients who are discharged to a nursing-home facility or receiving in-home rehabilitation by home care.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 169 (Actual)
Dates: Start 2021-04-06 (Actual); Primary Completion 2024-03-22 (Actual); Study Completion 2025-03-18 (Actual)

PRIMARY OUTCOMES:
Function in daily living (ADL). | Difference between groups at first follow up (6 weeks)
  For THA's: Hip disability and Osteoarthritis Outcome Score (HOOS) subscale: function in daily living (ADL).
  For TKA's: Knee injury and Osteoarthritis Outcome Score (KOOS) subscale: function in daily living (ADL).
  This subscale consists of 17 questions related to the patient's function in activities of daily living such as "descending stairs", "standing" and "getting in/out of car". The subscale is scored by the degree of difficulty the patient experiences in the last week on a 5-point Likert scale (none, mild, moderate, severe, and extreme), and calculated to a score ranging from 0 (worst/extreme difficulties) to 100 (best/ no problems). The total questionnaire takes about 10 minutes to complete. At least 50% of the questionnaire items are required to be answered to permit calculation of a mean score.

SECONDARY OUTCOMES:
Function in daily living (ADL) | Difference between groups at 3 and 12 months follow up.
  See above
Symptoms, pain and quality of life. | Baseline, 6 weeks, 3 and 12 months.
  For THA: 3 subscales in the patient-rapported questionnaire "HOOS" For TKA: 3 subscales in the patient-rapported questionnaire "KOOS".
  These subscales are scored by the degree of difficulty the patient has experienced in the last week on a 5-point Likert scale. Each subscale provides a score, which can be calculated to a total score ranging from 0 (worst/extreme difficulties) to 100 (best/ no problems). At least 50% of the questionnaire items in each subscale are required to be answered to permit calculation of a mean score.
Patient global assessment | Baseline, 6 weeks, 3 and 12 months.
  At baseline the patient's perception of his or her overall functional ability will be assessed using a single numeric rating scale, as recommended by OARSI. The patient will be asked a single question: "How would you rate your current level of function during your usual activities of daily living?" During follow-up assessment patients will be asked the same question as at baseline. Their answer will be rated on a 0-100 visual rating scale with end-points anchored as "Inability to perform any daily activities" (0) and "No problem with any daily activity" (100)
30-s chair stand test. | Baseline, follow up at 6 weeks, 3 and 12 months
  Performance-based assessment will be performed using the 30-s chair-stand test, which represent the sit-to-stand activity. The test counts the number of sit-to-stand repetitions the patient can perform in 30 seconds. The straight-back chairs used for testing during all outcome assessments will be of the same model, same height (approximately 43 cm), and will be placed against a wall. Any other adaptations (i.e. the use of armrests or assistive devices) will be reported. To assure understanding, two slow-paced repetitions will be practiced before the test initiates. The 30-s chair stand test has proven good reliability to measure functional performance following THA and TKA.
40 meters walking test. | Baseline, follow up at 6 weeks, 3 and 12 months
  This performance-based assessment measures short distance walking activity. The patient will be instructed to walk as quickly as safely as possible to a mark 10 meters away, return and repeat for a total distance of 40 meters. Each walk of 10 meters (excluding the turn time) is recorded and expressed as speed m/s by dividing distance by time in seconds. A practice walk up and back will be performed to assure understanding. Any assistive devices used will be recorded.
Use of analgesics | Baseline, follow up at 6 weeks, 3 and 12 months.
  The use of analgesics will recorded at baseline and at all follow-up assessments, using a nominal scale (yes/no) regarding the daily consumption of opioids, non-steroid-anti inflammatorily drug (NSAID) and paracetamol. If the patient were not aware of his or hers use of analgesics, a medical record will obtained to assess the use of analgesics.
Patient satisfaction | Follow up at 6 weeks.
  Patients will be asked to answer four questions to indicate their level of satisfaction. The answers will be based on a 4-Likert ordinal scale with the categories: very satisfied (100 points), somewhat satisfied (75 points), somewhat dissatisfied (50 points), and very dissatisfied (25 points). The score is the unweighted mean of the combined scores. The four questions are: "How satisfied are you with the results of your surgery and rehabilitation?", "How satisfied are you with your surgery and rehabilitation for improving your pain?", "How satisfied are you with the results of your surgery and rehabilitation for improving your ability to do home or yard work?" and "How satisfied are you with the results of surgery and rehabilitation for improving your ability to do recreational activities?". The questions are modified from the Self-Administered Patient Satisfaction Scale for Primary Hip and Knee Arthroplasty.
Time usage (care provider). | Baseline, follow up at 6 weeks, 3 and 12 months
  Analysis of the economical resources required for each of the three rehabilitation strategies. The principal investigator intend to use this data in a later cost-analysis.
Number of adverse events | Baseline, follow up at 6 weeks, 3 and 12 months
  Number and nature of adverse events during enrolment of the trial will be recorded, regardless of the relation to the trial.

OTHER OUTCOMES:
Homebased telerehabilitation + homebased rehabilitation group: Exercise adherence | Follow up at 6 weeks
  Exercise adherence will be measured as a percentage (0-100), where 0 % indicates total non-adherence and 100 % indicates total adherence to the exercise prescription. Exercise adherence is objectively recorded in the telerehabilitation group and can be extracted from the device used by the patients.

CONTACTS AND LOCATIONS:
Locations (1):
- Genoptræningen, Nørremøllecenteret, Nexø, Bornholm, Denmark

IPD SHARING:
Plan to Share IPD: Undecided